CLINICAL TRIAL: NCT05354349
Title: A Phase 1, Double-Blind, Placebo-Controlled, Single-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of PRA023 in Healthy Caucasian and Japanese Adult Volunteers
Brief Title: Bioavailability of SC Formulation and Japanese Ethnobridging Study for PRA023
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prometheus Biosciences, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: Altasciences Company Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PR200-105; 7240-004 (Other: Merck)
Record Dates: First submitted 2022-04-01; First posted 2022-04-29 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PRA023 SC/Placebo IV (Experimental): Participants randomized to receive active subcutaneous injection/placebo intravenous infusion
  Interventions: Drug: PRA023 SC; Drug: Placebo IV
- Placebo SC/PRA023 IV Low Dose (Active Comparator): Participants randomized to receive placebo subcutaneous injection/active intravenous infusion
  Interventions: Drug: PRA023 IV Low Dose; Drug: Placebo SC
- Placebo SC/Placebo IV (Placebo Comparator): Participants randomized to receive placebo subcutaneous injection/placebo intravenous infusion
  Interventions: Drug: Placebo IV; Drug: Placebo SC
- Placebo SC/PRA023 IV High Dose (Experimental)
  Interventions: Drug: Placebo SC; Drug: PRA023 IV High Dose

INTERVENTIONS:
Drug: PRA023 IV Low Dose — Drug
  Arms: Placebo SC/PRA023 IV Low Dose
Drug: PRA023 SC — Drug
  Arms: PRA023 SC/Placebo IV
Drug: Placebo IV — Placebo
  Arms: PRA023 SC/Placebo IV; Placebo SC/Placebo IV
Drug: Placebo SC — Placebo
  Arms: Placebo SC/PRA023 IV High Dose; Placebo SC/PRA023 IV Low Dose; Placebo SC/Placebo IV
Drug: PRA023 IV High Dose — Drug
  Arms: Placebo SC/PRA023 IV High Dose

SUMMARY:
This is a randomized double-blind, placebo-controlled, single-dose study to evaluate the safety, tolerability, and pharmacokinetics of PRA023 in healthy Caucasian and Japanese adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* Subjects are required to meet the following criteria in order to be included in the study:

  1. Japanese subjects must have both natural (not adopted) parents and four grandparents of Japanese origin.
  2. Caucasian subjects must be of European or Latin American descent (i.e., White).
  3. Male or female (of non-childbearing potential only) between minimum adult legal age (according to local laws for signing the informed consent document) and 55 years of age.
  4. Females must be of non-childbearing potential and must have undergone one of the following sterilization procedures, and have official documentation, at least 6 months prior to the first dose:

     1. hysteroscopic sterilization;
     2. bilateral tubal ligation or bilateral salpingectomy;
     3. hysterectomy;
     4. bilateral oophorectomy, or;
     5. be postmenopausal with amenorrhea for at least 1 year prior to the first dose and have FSH serum levels consistent with postmenopausal status as per Investigator judgment.
  5. Male subjects must use reliable forms of contraception during sexual intercourse with female partners from screening to 30 days after the end of dosing.
  6. Good general health as determined by medical history, and by results of physical examination, chest x-ray, vital signs, ECG, and clinical laboratory tests obtained within 28 days (4 weeks) prior to study drug administration.

Exclusion Criteria:

* Subjects with the following characteristics will be excluded from the study:

  1. History or presence of any clinically significant organ system disease that could interfere with the objectives of the study or the safety of the subjects.
  2. Blood pressure and heart rate are outside the ranges 90-140 mmHg systolic, 60-90mmHg diastolic, heart rate 60-100 beats/min.
  3. 12-lead ECG with any abnormality judged by the Investigator to be clinically significant, QRS >= 120 milliseconds (msec), or QTcF interval of > 450 msec for men or > 470msec for women.
  4. Presence or history of any abnormality or illness, which in the opinion of the Investigator may affect absorption, distribution, metabolism or elimination of the study drug.
  5. Any screening laboratory evaluation outside the laboratory reference range that is judged by the Investigator to be clinically significant.
  6. History of or current active tuberculosis (TB) infection; history of latent TB that has not been fully treated or current latent TB infection as indicated by a positive QuantiFERON-TB test.
  7. History of significant allergy to any medication as judged by the Investigator.
  8. History of alcohol or drug abuse within the past 24 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence, severity, causal relationship of treatment emergent adverse events | Up to 14 Weeks
F% in Caucasian subjects | Up to 10 Weeks
  Mean SC versus IV AUC(inf) values
Cmax in Japanese subjects | Up to 14 Weeks
  Maximum concentration after single dose
Tmax in Japanese subjects | Up to 14 Weeks
  Time to reach maximum concentration after single dose

SECONDARY OUTCOMES:
Cmax in Caucasian subjects | Up to 10 Weeks
  Maximum concentration after single dose
Tmax in Caucasian subjects | Up to 10 Weeks
  Time to reach maximum concentration after single dose
Immunogenicity rate | Up to 14 Weeks
Change in sTL1A levels | Up to 14 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prometheus Biosciences, Study Director — Clinicaltrials Call Center
Locations (1):
- Altasciences Clinical LA, Inc., Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/